CLINICAL TRIAL: NCT02849444
Title: Post-authorisation Observational Study for the Assessment of Renal Function Response to Treatment in Patients With Relapsed Multiple Myeloma and Creatinine Clearance <50 mL/Min/1.73 m2 (CrCl <50 mL/Min/1.73 m2)
Brief Title: A Study to Assess Renal Function Response to Treatment in Patients With Relapsed Multiple Myeloma and Creatinine Clearance
Acronym: MIR50
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CEL-MIE-2012-01
Record Dates: First submitted 2015-08-06; First posted 2016-07-29 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Multiple Myeloma
Keywords: renal function; Relapsed Multiple myeloma; anti-MM therapy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Moderate kidney failure: 30 ≤ CrCl < 50 mL/min/1.73 m2
  Interventions: Other: Anti-myeloma treatment at physician discretion
- Severe kidney failure: CrCl < 30 mL/min/1.73 m2
  Interventions: Other: Anti-myeloma treatment at physician discretion

INTERVENTIONS:
Other: Anti-myeloma treatment at physician discretion — non Interventional Study

SUMMARY:
A prospective, multicentre, post-authorisation observational study. The objective of this study is assess the response of renal function in clinical practice to anti-multiple myeloma therapy in patients with relapsed MM and CrCl <50 mL/min/1.73 m2.

DETAILED DESCRIPTION:
Prospective, multicentre, post-authorisation observational study. Study population: Patients with relapsed multiple myeloma and with CrCl <50 mL/min/1.73 m2, for whom the investigator decides to start a new line of anti-myeloma treatment as per normal clinical practice. The decision to prescribe treatment will be clearly disassociated from the decision to include the patient in the study.

300 patients are expected to be recruited (225 for Group 1 and 75 for Group 2) from 40 sites (approximately 7-8 patients for each site). Patients will be included consecutively in the study.

The inclusion will be stratified to ensure the presence of all stages of renal impairment (RI) in two groups:

Documentation of 300 patients is planned (a maximum of 225 in group 1 and a minimum of 75 in group 2) at 40 sites (approximately 7-8 patients per each site). The patients will be included in the study in a consecutive manner.

In order to ensure the correct stratification of the sample group a real time central registry will be kept for the patients included in each group. Once the required number of patients for one of the groups is completed, inclusion in that group will be closed at all sites, keeping inclusion for other groups open, and so on until the entire sample size is complete.

Primary objective: To assess the response of renal function in clinical practice to anti-multiple myeloma therapy in patients with relapsed MM and creatinine clearance <50 mL/min/1.73 m2 (CrCl <50 mL/min/1.73m2).

The prospective follow-up period will cover two phases:

1. Treatment phase: covers the entire time the patient is receiving the first anti-myeloma treatment for relapse* for which he/she is included in this study.
2. Follow-up phase: A 36-month extension period after the end of the first anti-myeloma treatment for relapse for which he/she was included in the study.

   * Any change in therapeutic regimens, for example, discontinuation or addition of a drug (except for changes in dose for some of the initial drugs) will mark the end of the treatment phase and the passing of the patient to the follow-up phase. In case of temporary interruptions in treatment under 30 days (or of any duration if the reason for interruption is toxicity) the patient will continue in the treatment phase, provided that the initial treatment regimen for the relapse it resumed.

Secondary objectives:

* To describe the clinical and demographic characteristics of patients with relapsed multiple myeloma and CrCl <50 mL/min/1.73 m2.
* To assess the response rate of renal function in clinical practice to anti-multiple myeloma therapy in patients with relapsed multiple myeloma and CrCl <50 mL/min/1.73 m2.
* To assess the response of renal function based on the therapeutic regimens administered.
* To explore the concordance of the kidney function response and that of the myeloma in the clinical practice to the anti-myeloma treatment between consecutive relapses in the same patient.
* To assess time-dependent response parameters.
* To analyse the safety of treatments administered in clinical practice.
* To describe the use of resources associated with anti-myeloma therapy in clinical practice that can be measured financially, and to explore the possible differences between the various therapeutic regimens administered.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both genders, aged equal or more than 18 years.
2. Patients with documented relapsed multiple myeloma according to International Myeloma Working Group ( IMWG) criteria.
3. Patients with documented renal damage defined as creatinine clearance <50 ml / min / 1.73 m2 (CrCl <50ml / min / 1.73m2).
4. Patients to whom the researcher decides to initiate anti-myeloma treatment for relapse with one or more agents according to clinical practice *.
5. Patients who consent in writing after it has been clearly explained to them the nature and purpose of the study (written informed consent).
6. Subject with any of the following characteristics (at least one of the 2 following options must be Yes):

   * Subjects who have not previously participated in the study
   * Subjects who have previously participated in the study, who meet all the inclusion criteria again and to whom none of the exclusion criteria apply, and whose current relapse is consecutive to the relapse that prompted their initial inclusion in the study.

     * The decision to prescribe treatment will be clearly dissociated from the decision to include the patient in the study

       * Clarification is provided as to the aim of the study, which is to encompass all relapse subcategories included in the International Myeloma Working Group consensus document published in 2006. Therefore, all patients with clinically relapsed multiple myeloma, who are in relapse following a complete response or in progression (including refractory cases) as defined in point 8.1 and in table 4 of the protocol, are considered eligible candidates for participation in the EPA-MIR 50 study, as long as they meet all the other criteria

Exclusion Criteria:

1. Patients who are participating in an interventional clinical trial * or who refuse to participate in the study.
2. Patients with CrCl <50 ml / min / 1.73m2 due to a cause other than multiple myeloma properly documented at the discretion of the investigator *.

   * The inclusion of patients who are participating in another observational study is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with relapsed /refractorymultiple myeloma and with CrCl <50 mL/min/1.73 m2, for whom the investigator decides to start a new line of anti-myeloma treatment as per normal clinical practice. The decision to prescribe treatment will be clearly disassociated from the decision to include the patient in the study.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2012-09-23 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Creatinine levels to determinates Renal function response | Up to 12 months
  Creatinine records from basal visit to last visit to determinates Creatinine clearance with the Cockcroft-Gault formula.
Age of participants at baseline to determinates Renal function response | Baseline visit
  Patient Age record to determinates Creatinine clearance with the Cockcroft-Gault formula.
Weight of participants at baseline to determinates Renal function response | Baseline visit
  Patient weight recorded in each visit to determinates Creatinine clearance with the Cockcroft-Gault formula.
Gender of participants at baseline to determinates Renal function response | Baseline visit
  Patient gender recorded in basal visit to determinates Creatinine clearance with the Cockcroft-Gault formula.

SECONDARY OUTCOMES:
Race of participants at Baseline | Baseline visit
  To describe the demographic characteristics of patients with relapsed multiple myeloma and CrCl <50 mL/min/1.73 m2.
Clinical Outcome of participants with Multiple Myeloma (MM) clinical description | Up to 12 months
  To describe the clinical characteristics of patients with relapsed multiple myeloma and CrCl <50 mL/min/1.73 m2.
Renal response rate assessment in clinical practice. | Up to 12 months
  Describe response rate of renal function according to eGFR and total proteinuria
Time dependent Renal response rate assessment in clinical practice. | Up to 12 months
  Time to best renal response
Type of Anti-myeloma therapeutic regimens. | Up to 12 months
  Describe various types of anti-myeloma regimens participants will receive.
Multiple Myeloma (MM) response to anti-myeloma treatment | Up to 12 months
  MM response evaluation according to IMWG criteria
MM response to Time to Progression | Up to 12 months
  Time to progression is defined as time from baseline to the appearance of the event; considering as an event progression or death from any cause.
MM response to Time to first response | Up to 12 months
  Time to response is defined as time from the date of the first dose of study treatment to the date of the first documented hematologic improvement.
MM response to Progression Free Survival | Up to 12 months
  Progression free survival is defined as time from the date of the first dose of study treatment to the date of the first documented disease progression or relapse per IWG 2006 criteria.
Adverse events (AEs) | Up to 12 months
  Number of participants with adverse events
Cost of visit to hospital/primary health care associated with anti-myeloma therapy | Up to 12 months
  To describe the costs associated with anti-myeloma therapy in clinical practice that can be measured financially, and to explore the possible differences between the various therapeutic regimens administered. This includes, visits to hospital/primary health care center.
Number of participants with relapsed kidney function | Up to 36 months
  Concordance of the kidney function response and that of the myeloma in the clinical practice to the anti-myeloma treatment between consecutive relapses in the same patient.

CONTACTS AND LOCATIONS:
Overall Officials: Mireya Navarro, MD, Study Director — Celgene Spain
Locations (40):
- Spain (40):
  - Hospital Torrecárdenas, Almería, Andalusia
  - Hospital Universitario Puerta del Mar, Cadiz, Andalusia
  - Hospital Virgen de la Nieves, Granada, Andalusia
  - Hospital Universitario Ciudad de Jaen, Jaén, Andalusia
  - Hospital general de jeréz, Jerez de la Frontera, Andalusia
  - Hospital Virgen de la macarena, Seville, Andalusia
  - Hospital Miguel Servet, Zaragoza, Aragon
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital de Insular de Gran Canaria, Las Palmas de Gran Canaria, Canary Islands
  - Hospital de Basurto, Bilbao, Castille and León
  - Hospital de Burgos, Burgos, Castille and León
  - Hospital de León, León, Castille and León
  - Rio Hortega de Valladolid, Valladolid, Castille and León
  - Hospital General de Ciudad Real, Ciudad Real, Castille-La Mancha
  - Hospital La Ribera, Alzira, Catalonia
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Vall d´Hebron, Barcelona, Catalonia
  - Hospital Clinic I Provincial de Barcelona, Barcelona, Catalonia
  - Hospital Duran reynls, Barcelona, Catalonia
  - Hospital Universitario Josep Trueta de Girona, Girona, Catalonia
  - Hospital Arnau de Vilanova de Lleida, Lleida, Catalonia
  - Hospital Sant Joan de manresa, Manresa, Catalonia
  - Hospital de Sabadell ( Parc Taulí), Sabadell, Catalonia
  - Hospital Mutua terrassa, Terrassa, Catalonia
  - Complejo Hospitalario Universitario Santiago, Santiago de Compostela, Galicia
  - Complejo Hospitalario Universitario de Vigo, Vigo, Galicia
  - Hospital san pedro, Logroño, La Rioja
  - Hospital Fundación de Alcorcón, Alcorcón, Madrid
  - Hospital Puerta de Hierro, Majadahonda, Madrid
  - Hospital Santa Lucía, Cartagena, Murcia
  - Hospital Virgen de Arrixaca, El Palmar, Murcia, Murcia
  - Hospital de Cabueñes, Gijón, Principality of Asturias
  - Hospital General de Alicante, Alicante, Valencia
  - Hospital Clínico Universitario Valencia, Valencia, Valencia
  - Hospital La fe, Valencia, Valencia
  - Hospital Gregorio marañon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Complejo Universitario de San Carlos, Madrid
  - Hospital Universitario La paz, Madrid
  - Hospital Dr peset, Valencia